CLINICAL TRIAL: NCT05490394
Title: Ambispective Cohort Study on the Correlation Between 4G/5G Polymorphism of Plasminogen Activator Inhibitor-1 (PAI-1) Promoter and Moderate to Severe Postoperative Acute Renal Injury in Patients With Aortic Dissection
Brief Title: Correlation Study of PAI-1 4G/5G Polymorphism and Postoperative AKI in Patients With Aortic Dissection
Status: Completed | Type: Observational
Sponsor: Xijing Hospital (Other)
Responsible Party: Principal Investigator, Chong Lei, MD & phD, Principal Investigator, Xijing Hospital
Other Study IDs: KY20212193-F-1
Record Dates: First submitted 2022-08-03; First posted 2022-08-05 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-02

CONDITIONS: AKI - Acute Kidney Injury; PAI-1 4G/5G Polymorphism; Aortic Dissection
MeSH Terms: conditions — Acute Kidney Injury; Aortic Dissection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To explore the association between PAI-1 4G5G polymorphism and the risk of CSA-AKI in Stanford type A dissection patients undergoing open-heart repair surgery.

DETAILED DESCRIPTION:
The incidence of postoperative acute kidney injury（AKI）after cardiac surgery is high, especially in patients with aortic dissection. Moderate to severe postoperative AKI (stage 2 and 3 AKI) is closely related to the poor prognosis after cardiac surgery. Patients with Stanford type A dissection who suffered from stage 2 and 3 postoperative AKI will have a 4.45 times higher mortality than that of patients without AKI. At present, there is no effective treatment for cardiac surgery associated AKI (CSA-AKI), and prevention is more important than treatment. Therefore, screening high-risk patients and implementing individualized preventive measures are of great significance for the prevention of postoperative AKI and improvement of prognosis of patients.

The previous completed RCT study in the investigators' center showed that perioperative administration of inhaled nitric oxide (NO) to patients undergoing cardiopulmonary bypass (CPB) assisted multivalve replacement surgery could significantly reduce the incidence of postoperative AKI, but the NO should be provided before CPB was started, that is, when injury began. This phenomenon implied that NO played a preventive role rather than a therapeutic role. In further studies, the investigators found that the kidney protective mechanism of NO inhalation may be related to its role on PAI-1 regulation. According to the literature, the 4G5G polymorphism in the promoter region of PAI-1 is a natural regulator of the expression level of PAI-1 in vivo. Based on these findings, the investigators reviewed some cases who underwent aortic dissection correction surgery and also PAI-1 4G5G polymorphism test in our hospital, the investigators found that 4G/4G homozygous patients had a much higher proportion of moderate to severe AKI than 4G5G heterozygous patients or 5G/5G homozygous patients. However, due to the small sample size, the differences in AKI incidence between different genotype groups were not statistical significant.

In order to further explore the association between PAI-1 4G5G polymorphism and the risk of CSA-AKI, the investigators planed to expand the sample size and form a ambispective cohort study which include the retrospective cohort mentioned above and a new prospective cohort study. A total of 255 patients will be included to determine the genetic susceptibility of CSA-AKI associated with PAI-1 4G5G deletion / insertion polymorphism. All subjects included in the prospective part of this study will receive PAI-1 4G5G polymorphism test, and record whether postoperative AKI occurs and also AKI stage. There is no other intervention for patients included in this study in addition to blood collection. All medical decision-making processes in hospital will not be interfered by the research.

ELIGIBILITY:
Inclusion Criteria:

* Stanford type A aortic dissection patient admitted to the Department of Cardiology, in Xijing Hospital
* Open thoracic aortic dissection correction (total aortic arch replacement with or without aortic valve replacement) is proposed
* Age ≥ 18 years old
* Informed consent has been signed

Exclusion Criteria:

* Cardiopulmonary bypass assisted cardiac surgery has been performed in the past three months
* Renal failure patients who have started or are receiving dialysis treatment before operation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: For retrospective cohort: patients who previously underwent open thoracic aortic dissection correction surgery and also underwent PAI-1 4G5G polymorphism in Xijing Hospital.
  For prospective cohort: patients who is scheduled for open thoracic aortic dissection correction surgery (total aortic arch replacement, with or without aortic valve replacement) in Xijing Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 283 (Actual)
Dates: Start 2022-04-28 (Actual); Primary Completion 2022-06-16 (Actual); Study Completion 2022-08-01 (Actual)

PRIMARY OUTCOMES:
Number of participants who develop postoperative moderate to severe AKI | from time of the end of surgery; assessed up to 7 days
  number of participants who develop stage 2 to stage 3 AKI after the surgery

SECONDARY OUTCOMES:
Number of participants who develop postoperative AKI | from time of the end of surgery; assessed up to 7 days
  number of participants who develop all stage AKI after the surgery
In-hospital mortality | from time of the end of surgery; assessed up to 7 days
  incidence of deaths happened after surgery during the hospital stay
Length of stay in hospital | from time of the end of surgery; assessed up to 7 days
  duration of postoperative stay in hospital

CONTACTS AND LOCATIONS:
Locations (1):
- Xijing Hospital, Xi'an, Shaanxi, China